CLINICAL TRIAL: NCT01204996
Title: An Open-label, Multicenter, Phase 1b Study of CNTO 888 (an Anti-CCL 2 Monoclonal Antibody) in Combination With Chemotherapies for the Treatment of Subjects With Solid Tumors
Brief Title: A Study of the Safety and Efficacy of CNTO 888 in Combination With SoC (Standard of Care) Chemotherapy in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sr. Director, Clinical Leader, Centocor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016462; 2009-015541-23 (EudraCT Number); CNTO888STM1002 (Other: Centocor)
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Cancer
Keywords: monoclonal antibody; solid tumor; chemotherapy; standard of care
MeSH Terms: conditions — Neoplasms | interventions — carlumab; Gemcitabine; Paclitaxel; Carboplatin; Docetaxel

ARMS (4):
- 1 (Experimental): CNTO888 + docetaxel 15 mg/kg CNTO 888 every 3 weeks plus docetaxel 75 mg/m2 every 3 weeks
  Interventions: Drug: CNTO888 + docetaxel
- 2 (Experimental): CNTO888 + gemcitabine 15 mg/kg CNTO 888 every 3 weeks plus gemcitabine 1000 mg/m2 administered on Days 1 and 8 of the 3-week cycle
  Interventions: Drug: CNTO888 + gemcitabine
- 3 (Experimental): CNTO888 + Paclitaxel and carboplatin 15 mg/kg CNTO 888 every 3 weeks plus paclitaxel 175 mg/m2 and carboplatin dosed to AUC 6 every 3 weeks
  Interventions: Drug: CNTO888 + Paclitaxel and carboplatin
- 4 (Experimental): CNTO888+DOXIL®/ Caelyx® doxorubicin HCl liposome injection 10 mg/kg CNTO 888 every 2 weeks plus DOXIL®/Caelyx® (doxorubicin HCl liposome injection) 50 mg/m2 every 4 weeks
  Interventions: Drug: CNTO888+DOXIL®/ Caelyx® doxorubicin HCl liposome injection

INTERVENTIONS:
Drug: CNTO888+DOXIL®/ Caelyx® doxorubicin HCl liposome injection — 10 mg/kg CNTO 888 every 2 weeks plus DOXIL®/Caelyx® (doxorubicin HCl liposome injection) 50 mg/m2 every 4 weeks
  Arms: 4
Drug: CNTO888 + gemcitabine — 15 mg/kg CNTO 888 every 3 weeks plus gemcitabine 1000 mg/m2 administered on Days 1 and 8 of the 3-week cycle
  Arms: 2
Drug: CNTO888 + Paclitaxel and carboplatin — 15 mg/kg CNTO 888 every 3 weeks plus paclitaxel 175 mg/m2 and carboplatin dosed to AUC 6 every 3 weeks
  Arms: 3
Drug: CNTO888 + docetaxel — 15 mg/kg CNTO 888 every 3 weeks plus docetaxel 75 mg/m2 every 3 weeks
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and dose regimen of CNTO 888 when administered to patients with solid tumors in combination with 4 standard of care chemotherapy regimens.

DETAILED DESCRIPTION:
CNTO 888 is an antibody that works by blocking a protein called CC-chemokine ligand 2 (CCL2). In research studies CCL2, has been shown to increase the growth of new blood vessels which help the tumor to survive. It is hoped that blocking CCL2 may help to control tumor growth.

Patients will receive one of four treatments. A dose of 15 mg/kg CNTO 888 will be administered once every 3 weeks in combination with either docetaxel, gemcitabine, or paclitaxel-carboplatin in Treatment Arms 1, 2, and 3, respectively; and 10 mg/kg CNTO 888 will be administered once every 2 weeks with DOXIL® / Caelyx® (doxorubicin HCl liposome injection) for intravenous infusion once every 4 weeks in Treatment Arm 4. The maximum time that patients will be in the study is one year.

Safety assessments will be conducted throughout the course of the study. Safety assessments include the monitoring of side effects,clinical laboratory tests (hematology, biochemistry, and urinalysis), vital signs, and physical examinations. CNTO 888 will be administered IV at 2 different doses (15 mg/kg or 10 mg/kg) dependant on the chemotherapy combination. Combination therapy will be continued until disease progression, unacceptable toxicity, the patient refuses further combination therapy, withdraws consent, or is treated for 1 year

ELIGIBILITY:
Inclusion Criteria:

* Documentation of an advanced solid tumor
* No more than 2 previous anticancer therapies
* good performance status
* adequate bone marrow, liver, and renal function / adequate blood test values
* willing to use birth control measures

Exclusion Criteria:

* No residual toxicities resulting from previous therapy
* no known allergies, hypersensitivity, or intolerance to antibodies or chemotherapies
* clinically significant bleeding or requiring concurrent therapeutic dose of anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-05; Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the safety of CNTO 888 when administered to patients with solid tumors in combination with 4 standard of care chemotherapy regimens. | During treatment and up to 30 days after last study treatment

SECONDARY OUTCOMES:
Pharmacokinetics(rate of movement in the body and then the clearance) | during study as specified in the protocol (interim analysis) and at End of Study (1 year)
Pharmacodynamics (action of drug on body systems) | during study as specified in the protocol (interim analysis) and at End of Study (1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (5):
- United States (2):
  - Detroit, Michigan
  - Tacoma, Washington
- Spain (3):
  - Barcelona
  - Madrid
  - PAU de Sanchinarro

REFERENCES:
- [Derived] Brana I, Calles A, LoRusso PM, Yee LK, Puchalski TA, Seetharam S, Zhong B, de Boer CJ, Tabernero J, Calvo E. Carlumab, an anti-C-C chemokine ligand 2 monoclonal antibody, in combination with four chemotherapy regimens for the treatment of patients with solid tumors: an open-label, multicenter phase 1b study. Target Oncol. 2015 Mar;10(1):111-23. doi: 10.1007/s11523-014-0320-2. Epub 2014 Jun 15. PMID 24928772